CLINICAL TRIAL: NCT02952404
Title: Incidence of Obstetric Anal Sphincter Injuries After Training to Protect the Perineum
Brief Title: Incidence of Obstetric Anal Sphincter Injuries After a Protection Training
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 15-050
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Obstetric Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before workshop: October 2014 to October 2015 Cohort which is the time frame before the educational workshop
- After workshop: December 2015 to December 2016 Cohort which is the time after the educational workshop
  Interventions: Procedure: Educational workshop

INTERVENTIONS:
Procedure: Educational workshop — The educational workshop for improved perineal support during vaginal delivery
  Groups: After workshop

SUMMARY:
This is a retrospective cohort study. This two cohort study seeks to compare the incidence of obstetric anal sphincter injuries (OASIS) in two time periods, before and after an educational workshop for improved perineal support.

DETAILED DESCRIPTION:
Perineal trauma during vaginal delivery is a major health issue associated with significant morbidity. It has been associated with many long term sequelae, including urinary and fecal incontinence. Specifically, third and fourth degree lacerations are known risk factors for the development of fecal incontinence.

Due to their serious impact, third or fourth degree perineal tears are a commonly tracked adverse event in obstetric care (Agency for Healthcare Research and Quality and Joint Commission). As such, incidence data will soon be available to third-party payers and to the public on the Internet. Moreover, functional impairment after perineal lacerations continues to be a significant impetus for legal claims. Thus, reducing OASIS while preserving maternal and fetal outcomes is an important goal in clinical obstetrics.

At the two TriHealth tertiary care institutions, the overall rate of OASIS is 3.5%. This is comparable, but not superior, to published rates at other centers. In fact, the literature is quite variable, with reported incidences ranging from 0.25-6%. Indeed, TriHealth has recently set up a task force to reduce these injuries as part of recent endeavors for quality improvement. Prevention is the first step in improving these complications.

This study seeks to decrease the incidence of obstetric and anal sphincter injuries that may occur during the birthing process by bringing in a notable physician to review techniques with the obstetrics residents to help avoid these injuries then observe the deliveries of the women enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Obstetrics resident patients
* 18 years and older women who delivered vaginally between Oct. 2014 and Dec.2016

Exclusion Criteria:

* Women who delivered by cesarean section, preterm deliveries (less than 32 weeks), and multiple gestations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Resident patients, 18 years and older women, who delivered vaginally between October 2014 and December 2016.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Incidence of obstetric anal sphincter injuries | before (between Oct. 2014 and Oct. 2015) and after (between Dec. 2015 and Dec. 2016_) an educational workshop (Nov. 2015)
  This is identified by ICD-9 code of third or fourth degree lacerations.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No